CLINICAL TRIAL: NCT00754611
Title: The Evolution and Management of Migraine Recurrence Beyond 24 Hours: A Prospective Study of Tertiary Care Center Patients
Brief Title: The Evolution and Management of Migraine Recurrence Beyond 24 Hours
Status: Completed | Type: Observational
Sponsor: Rowan University (Other)
Collaborators: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: EN4162008
Record Dates: First submitted 2008-09-09; First posted 2008-09-18 (Estimated); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
What is the course of migraine headache recurrence, how is it managed, what characteristics are associated with it, and how does it influence patient satisfaction with treatment?

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients at University Headache Center with > 6 month diagnosis of migraine with and/or without aura (ICHD-II)
* Greater than or equal to 18 years old

Exclusion Criteria:

* Greater than 15 days/month total headache days
* Analgesic use greater than 15 days/month (other than aspirin less than or equal to 325mg/d)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at the University Headache Center, aged 18 or older, with a diagnosis of migraine with and/or without aura as defined by ICHD-II criteria
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Primary efficacy outcomes will be sustained pain free response between 4 and 72 hours after initial abortive medication dosing (lack of recurrence over 72 hours) | 4 to 72 hours

SECONDARY OUTCOMES:
Pain response and pain free data | 30 minutes, 1,2,4,24,48,and 72 hours
Rate of recurrence, time of recurrence, time to re-dosing | 72 hours
Rate of recurrence among multiple attacks per subject | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Loretta Mueller, DO, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- University of Medicine and Dentistry of New Jersey, Stratford, New Jersey, United States